CLINICAL TRIAL: NCT01653353
Title: Swiss Study on Vitamin D and Calcium in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SSVDNH
Record Dates: First submitted 2012-07-23; First posted 2012-07-31 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: Aging; Vitamin Deficiency
Keywords: nursing home; vitamin D supplements; calcium supplements; guideline adherence
MeSH Terms: conditions — Avitaminosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Entire group (Experimental): A peer-applied guideline will be applied to the physicians.
  Interventions: Behavioral: peer physician-applied recommendation to the physicians

INTERVENTIONS:
Behavioral: peer physician-applied recommendation to the physicians — The peer physician-applied recommendation will include scientific information, practical recommendations to correctly supplement with calcium and vitamin D and a list of individual appraisals of the prescribed supplements among the residents.

SUMMARY:
Residents of nursing homes are endangered by malnutrition and vitamin D deficiency. Our study checks compliance with Swiss federal recommendations on vitamin D and calcium supplementation among residents of a Swiss nursing home. A peer physician-applied recommendation on compliance with the federal recommendations with individual evaluation of the residents will be sent to the physicians in care. After one year, data will be collected again.

DETAILED DESCRIPTION:
The investigators plan to get a complete sample of all inhabitants, so the only inclusion criterion is to get an informed consent either from the residents or from their relatives. The following data will be recorded: Year of birth, gender, height, weight, blood pressure and heart rate, daily calcium intake from diet, nursing home scales on pain, depression, dementia and activities of daily life, date of entry to the home, diagnosis and medication lists. From a venous blood sample the investigators get: calcium, phosphate, albumin, creatinin, 25-hydroxyvitamin D, parathormone (intact).

Primary endpoint: Proportion of medication lists of residents complying with federal recommendation on vitamin D and calcium supplementation.

Secondary endpoints: 25-hydroxyvitamin D levels, effect of an intervention with a nursing home-applied recommendation to the physicians.

ELIGIBILITY:
Inclusion Criteria:

* Resident of nursing home on qualifying date
* Written informed consent by residents or their relatives

Exclusion Criteria:

* Refusion of participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Proportion of compliance with federal recommendations | up to 12 months
  We register the proportion of residents those calcium and vitamin D supplementation complies with Swiss federal recommendation.

SECONDARY OUTCOMES:
25-hydroxyvitamin D serum levels | up to 12 months
  We measure 25-hydroxyvitamin D serum levels among the residents.
Effect of nursing home-applied recommendations to physicians | up to 12 months
  We check the effect of a nursing-home-applied recommendation to the physicians in care of the residents concerning correct supplementation with vitamin D and calcium on a) proportion of compliance with federal recommendations, b) 25-hydroxyvitamin D serum levels and c) medication costs.

CONTACTS AND LOCATIONS:
Overall Officials: Markus P. Gnädinger, MD, Principal Investigator — University of Zurich; Heike A. Bischoff-Ferrari, MD, DrPH, Prof, Study Director — University of Zurich; Andreas Egli, MD, Study Chair — University of Zurich
Locations (1):
- Pflegeheim Sonnhalden, Arbon, Thurgau, Switzerland